CLINICAL TRIAL: NCT00110994
Title: Phase II Randomized, Placebo Controlled Study of Sorafenib in Repeated Cycles of 21 Days in Combination With Dacarbazine (DTIC) Chemotherapy in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Treatment for Subjects With Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11715
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Cancer; Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Sorafenib; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + Dacarbazine (Experimental): Sorafenib, 2 tablets (200 mg each) orally twice daily (bid) on study days 1-21 + Dacarbazine, 1000 mg/m^2 intravenous on study day 1 (21 days per cycle) for double-blind (DB) treatment. Subjects who discontinued DB treatment with complete response (CR), partial response (PR) or stable disease (SD) entered active follow up period. Subjects who discontinued DB treatment with disease progression (DP) entered long term follow up period.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Dacarbazine
- Placebo + Dacarbazine (Active Comparator): Placebo, 2 tablets orally twice daily on study days 1-21 + Dacarbazine, 1000 mg/m^2 intravenous on study day 1 (21 days per cycle) for double-blind (DB) treatment. Subjects who discontinued DB treatment with complete response (CR), partial response (PR) or stable disease (SD) entered active follow up period. Subjects who discontinued DB treatment with disease progression (DP) entered long term follow up period.
  Interventions: Drug: Placebo; Drug: Dacarbazine

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib, 400 mg, 2 tablets (200 mg each) po (per os) bid (twice daily) Study days 1-21
  Arms: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine
Drug: Placebo — Placebo, 2 tablets, po (per os) bid (twice daily) Study days 1-21
  Arms: Placebo + Dacarbazine
Drug: Dacarbazine — Dacarbazine, 1000 mg/m^2 intravenous on Study Day 1

SUMMARY:
This is a randomized, double blind, placebo controlled, multicenter, phase II study to compare the anti-tumor activity as measured by progression-free survival (PFS) and the tolerability of Sorafenib in combination with Dacarbazine (DTIC) versus DTIC in combination with placebo in subjects with unresectable Stage III or Stage IV melanoma who have not received prior cytotoxic chemotherapy. A total of approximately 98 subjects will be randomized to receive DTIC + Sorafenib or DTIC + Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a life expectancy of at least 12 weeks
* Patients with histologically or cytologically confirmed unresectable (Stage III) or metastatic (Stage IV) melanoma
* Patients who have an ECOG PS of 0, or 1
* Measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST criteria

Exclusion Criteria:

* Primary ocular or mucosal melanoma
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta [Noninvasive papillary carcinoma], Tis [Carcinoma in situ: "flat tumor"] & T1 [Tumor invades subepithelial connective tissue]) or any cancer curatively treated < 3 years prior to study entry
* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- United States (12):
  - Tucson, Arizona
  - Aurora, Colorado
  - Lakeland, Florida
  - Park Ridge, Illinois
  - Boston, Massachusetts
  - St Louis, Missouri
  - Omaha, Nebraska
  - Charlotte, North Carolina
  - Pittsburgh, Pennsylvania
  - Hilton Head Island, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas

REFERENCES:
- [Result] McDermott DF, Sosman JA, Gonzalez R, Hodi FS, Linette GP, Richards J, Jakub JW, Beeram M, Tarantolo S, Agarwala S, Frenette G, Puzanov I, Cranmer L, Lewis K, Kirkwood J, White JM, Xia C, Patel K, Hersh E. Double-blind randomized phase II study of the combination of sorafenib and dacarbazine in patients with advanced melanoma: a report from the 11715 Study Group. J Clin Oncol. 2008 May 1;26(13):2178-85. doi: 10.1200/JCO.2007.14.8288. PMID 18445842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 121 subjects were enrolled at 17 centers in the United States. There were 20 screening failures; 12 subjects did not meet 1 or more entry criteria, 4 subjects withdrew consent before randomization, and 4 subjects were not randomized for other reasons. 101 subjects were randomized between 21 Mar 2005 and 27 Apr 2006.
Pre-assignment Details: A total of 101 subjects were randomized (50 to Placebo + Dacarbazine (DTIC) and 51 to Sorafenib + DTIC) and were included in the population valid for intent to treat (ITT) analyses. All randomized subjects received study drug and were included in the population valid for safety analyses.
Period: Double-blind (DB) Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Started | 51 (ITT population) | 50 (ITT population)
Received Treatment | 51 (Safety population) | 50 (Safety population)
Completed | 9 | 3
Not Completed | 42 | 47
Not completed — Adverse Event | 3 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Progression by clinical judgement | 2 | 1
Not completed — Radiological and symptomatic progression | 34 | 41
Not completed — other reasons | 2 | 3
Period: Active Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Started | 1 (Subjects discontinued DB treatment with CR, PR and SD entered this period.) | 2 (Subjects discontinued DB treatment with CR, PR and SD entered this period.)
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Disease progression/recurrence/replace | 1 | 0
Not completed — Other reasons | 0 | 2
Period: Long Term Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Started | 41 (Subjects discontinued DB treatment with DP entered this period.) | 47 (Subjects discontinued DB treatment with DP entered this period.)
Completed | 22 | 30
Not Completed | 19 | 17
Not completed — Death | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.7) | 60.1 (13.8) | 58.3 (13.3)
Age, Customized [Number; unit: participants]
  <65 years | 36 | 33 | 69
  >=65 and <75 years | 11 | 8 | 19
  >=75 years | 4 | 9 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 38 | 33 | 71
American Joint Committee on Cancer (AJCC) Stage at Study Entry [Number; unit: participants] — Stage III: Clinical or radiological evidence of regional metastases (M), in either the lymph nodes or intra-lymphatic. Stage IV: M at any distant site. M1a: M to the skin, subcutaneous tissue, or lymph nodes. M1b: M to the lung. M1c: M to all other visceral sites or at any site associated with an elevated serum lactate dehydrogenase.
  participants
    Stage III | 2 | 1 | 3
    Stage IV M1a | 3 | 7 | 10
    Stage IV M1b | 18 | 17 | 35
    Stage IV M1c | 28 | 25 | 53
Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). Subjects entering this study must have had an ECOG score of 0 or 1 (restricted in physically strenuous activity but ambulatory).
  participants
    Status 0 | 31 | 31 | 62
    Status 1 | 20 | 19 | 39
Lactate dehydrogenase (LDH) at study entry [Number; unit: participants] — Lactate dehydrogenase (LDH) was assessed at study entry as part of a battery of tests to assess liver function. A typical normal range is 105 to 333 Units/Liter (U/L), but may vary across laboratories.
  participants
    Normal | 33 | 29 | 62
    Low | 1 | 2 | 3
    High | 12 | 17 | 29
    Missing | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated as the time (days) from date of randomization to date of first observed DP (per modified Response Evaluation Criteria In Solid Tumors [RECIST] or clinical judgment, whichever was earlier: CR, PR, stable disease, progressive disease) or death due to any cause, if death occurred before progression was documented. The actual date of tumor assessments was used for this calculation. PFS for subjects without progression or death was censored at the last date of tumor evaluation. PFS for subjects who had no tumor assessments after baseline and did not die was censored at 1 day.
Time Frame: Time from randomization to documented tumor progression or death (the maximum treatment duration of 71.1 weeks)
Population: PFS was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
days | 148 [112 to 196] | 82 [43 to 125]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.068, log rank test; Hazard Ratio (HR) = 0.665, 95% CI 2-sided [0.428 to 1.034]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was calculated as the number of days from date of randomization to death date. Subjects who had not died at the time of analysis were censored at their last contact date.
Time Frame: Time from randomization to death (the maximum treatment duration of 71.1 weeks)
Population: OS was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
days | 319 [245 to 492] | 359 [285 to 504]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.973, log rank test; Hazard Ratio (HR) = 0.992, 95% CI 2-sided [0.627 to 1.570]

3. Secondary Outcome: Number of Participants in Tumor Response Categories
Description: Tumor response was defined as the best response (confirmed complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD]) assessed using the Response Evaluation Criteria in Solid Tumors (RECIST). PR: At least a 30% decrease in the sum of the longest diameter [SLD] of target lesions, taking as reference the baseline SLD. CR: Disappearance of all target lesions. SD: Does not qualify for CR or PR. PD: at least a 20% increase in SLD taking as reference the smallest SLD recorded since treatment started or the appearance of one or more new lesions.
Time Frame: Every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: Tumor response was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
participants
  CR | 0 | 0
  PR | 12 | 6
  SD | 24 | 22
  PD | 15 | 21
  Not Evaluated | 0 | 1

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was calculated as the time (days) from date of randomization to date of first observed disease progression (per modified RECIST or clinical judgment, whichever was earlier: CR, PR, stable disease, progressive disease). The actual dates of tumor assessments were used for this calculation. TTP for subjects without disease progression at the time of analysis, including subjects with death prior to progression, was censored at the last date of tumor evaluation. TTP for subjects who had no tumor assessments after baseline was censored at 1 day.
Time Frame: Time from randomization to documented tumor progression (median time of 148 days)
Population: TTP was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
days | 148 [112 to 199] | 82 [43 to 125]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.039, log rank test; Hazard Ratio (HR) = 0.619, 95% CI 2-sided [0.391 to 0.980]

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from the first documented objective response of Partial Response (PR: At least a 30% decrease in the sum of the longest diameter [SLD] of target lesions, taking as reference the baseline SLD or better) or Complete Response (CR: Disappearance of all target lesions), whichever was noted earlier, to disease progression or death (if death occurred before progression was documented). Duration of response for subjects who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment.
Time Frame: Time from initial response to documented tumor progression or death (median time of 188 days)
Population: DOR was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
days | 188 [144 to 252] | 161 [126 to 203]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.194, log rank test; Hazard Ratio (HR) = 0.427, 95% CI 2-sided [0.114 to 1.601]

6. Secondary Outcome: Change in Eastern Cooperative Oncology Group (ECOG) Performance Status From Baseline to the Visit When the Best Tumor Response Was Noted
Description: Change in ECOG PS is defined as an improvement (increase) or worsening (decrease) of at least one grade from the baseline ECOG score (from 0 [fully active] to 5 [dead]). Change in ECOG PS was recorded at the visit at which best confirmed response (BCR) using the modified RECIST (PR, CR, stable disease or Progressive Disease (PD)) was first noted (the change was 7% for both Sorafenib and Placebo). The BCR is the BCR recorded from the start of the treatment until DP/recurrence (taking as reference for DP, the smallest measurements recorded since treatment started).
Time Frame: Baseline and every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: Change in ECOG performance status was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
participants
  missing | 1 | 1
  better | 1 | 2
  no change | 34 | 34
  worse | 15 | 13

7. Secondary Outcome: Change of European Quality of Life 5-dimensional (EQ-5D) Questionnaire Index Score From Baseline to the Visit at Which Best Response Was First Noted
Description: European Quality of Life 5-dimensional (EQ-5D) is a self-administered questionnaire developed to measure health status across 5 dimensions: Mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension has 3 levels of response: No problem (1), some problems (2), and extreme problems (3). The five dimensions are summarized into a single score, the EQ-5D index score, which ranges between 0 and 1, with 0 representing the worst imaginable health state or death and 1 representing perfect health.
Time Frame: Baseline and every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: Change of EQ-5D questionnaire index score was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
scores on a scale | -0.004 (0.142) | -0.008 (0.125)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.908, t-test, 2 sided

8. Secondary Outcome: Change of European Quality of Life 5-dimensional (EQ-5D) Questionnaire Index Score From Baseline to the End of Treatment
Description: as for outcome 7
Time Frame: Baseline and every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
scores on a scale | -0.015 (0.124) | -0.019 (0.161)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.890, t-test, 2 sided

9. Secondary Outcome: Change of European Quality of Life Visual Analogue Scale (EQ-VAS) Score From Baseline to the Visit at Which Best Response Was First Noted
Description: European Quality of Life Visual Analogue Scale (EQ-VAS) is a self-administered test that records the respondents' self-rated health status on a visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). Responders specify their scales by indicating a position along a continuous line between 0 and 100.
Time Frame: Baseline and every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: Change of EQ-VAS score was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
scores on a scale | 0.558 (17.86) | -4.425 (17.28)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.201, t-test, 2 sided

10. Secondary Outcome: Change of European Quality of Life Visual Analogue Scale (EQ-VAS) Score From Baseline to the End of Treatment
Description: as for outcome 9
Time Frame: Baseline and every 6 weeks from the start of the treatment until the end of treatment visit with a median of 134 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Number analyzed (Participants) | 51 | 50
scores on a scale | -2.00 (19.612) | -8.146 (20.905)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Dacarbazine vs Placebo + Dacarbazine; Test type: Superiority or Other; p = 0.168, t-test, 2 sided

ADVERSE EVENTS:
Description: Abbreviations used in the Adverse Events section: Absolute Neutrophil Count (ANC), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Central Nervous System (CNS), Common Terminology Criteria for Adverse Events (CTCAE), Gastro-Intestinal (GI), National Cancer Institute (NCI), Not Otherwise Specified (NOS)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine | Placebo + Dacarbazine
Serious Adverse Events (participants affected / at risk) | 22/51 | 14/50
Other Adverse Events (participants affected / at risk) | 49/51 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine (N=51) | Placebo + Dacarbazine (N=50)
platelets (Blood and lymphatic system disorders) | 1 | 1
neutrophils (Blood and lymphatic system disorders) | 0 | 1
hemoglobin (Blood and lymphatic system disorders) | 0 | 1
leukocytes (Blood and lymphatic system disorders) | 1 | 0
supraventricular arrhythmia, atrial fibrillation (Cardiac disorders) | 1 | 0
supraventricular arrhythmia, supraventricular tachycardia (Cardiac disorders) | 0 | 1
hypotension (Cardiac disorders) | 4 | 0
cardiac ischemia / infarction (Cardiac disorders) | 2 | 0
cardiopulmonary arrest (Cardiac disorders) | 0 | 1
hypertension (Cardiac disorders) | 1 | 0
death not associated with CTCAE term, disease progression NOS (General disorders) | 2 | 1
death not associated with CTCAE term, multi-organ failure (General disorders) | 1 | 0
fever (General disorders) | 2 | 1
constitutional symptoms - other (General disorders) | 1 | 2
rigors / chills (General disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 3 | 1
nausea (Gastrointestinal disorders) | 2 | 1
ascites (Gastrointestinal disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1
dehydration (Gastrointestinal disorders) | 0 | 1
CNS hemorrhage (Vascular disorders) | 4 | 0
hemorrhage, GI, abdomen NOS (Vascular disorders) | 1 | 0
hemorrhage, GI, upper GI NOS (Vascular disorders) | 0 | 1
hemorrhage - other (Vascular disorders) | 1 | 0
hemorrhage pulmonary, nose (Vascular disorders) | 0 | 1
cholecystitis (Hepatobiliary disorders) | 2 | 0
liver dysfunction (Hepatobiliary disorders) | 1 | 0
pancreatitis (Hepatobiliary disorders) | 1 | 0
infection - other (Infections and infestations) | 1 | 1
infection with unknown ANC, skin (cellulitis) (Infections and infestations) | 0 | 1
fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
CNS ischemia (Nervous system disorders) | 0 | 1
dizziness (Nervous system disorders) | 1 | 0
neurology - other (Nervous system disorders) | 1 | 0
psychosis (Nervous system disorders) | 0 | 1
seizure (Nervous system disorders) | 0 | 1
blurred vision (Eye disorders) | 1 | 0
pain, chest / thorax NOS (General disorders) | 1 | 1
pain, abdomen NOS (General disorders) | 1 | 1
pain, extremity - limb (General disorders) | 0 | 1
pain, head / headache (General disorders) | 1 | 0
pain, muscle (General disorders) | 0 | 1
pain, pain NOS (General disorders) | 1 | 0
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
renal failure (Renal and urinary disorders) | 2 | 0
renal - other (Renal and urinary disorders) | 1 | 0
thrombosis / thrombus / embolism (Vascular disorders) | 2 | 0
no code in CTCAE (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Dacarbazine (N=51) | Placebo + Dacarbazine (N=50)
allergic reaction (Immune system disorders) | 3 | 0
platelets (Blood and lymphatic system disorders) | 30 | 14
neutrophils (Blood and lymphatic system disorders) | 23 | 9
hemoglobin (Blood and lymphatic system disorders) | 18 | 12
leukocytes (Blood and lymphatic system disorders) | 13 | 7
lymphopenia (Blood and lymphatic system disorders) | 3 | 1
hypertension (Cardiac disorders) | 5 | 0
hypotension (Cardiac disorders) | 4 | 0
fatigue (General disorders) | 29 | 27
weight loss (General disorders) | 9 | 4
rigors / chills (General disorders) | 5 | 3
sweating (General disorders) | 5 | 2
fever (General disorders) | 2 | 3
nausea (Gastrointestinal disorders) | 29 | 26
diarrhea (Gastrointestinal disorders) | 29 | 8
anorexia (Gastrointestinal disorders) | 17 | 11
vomiting (Gastrointestinal disorders) | 15 | 8
constipation (Gastrointestinal disorders) | 8 | 12
heartburn (Gastrointestinal disorders) | 5 | 5
GI - other (Gastrointestinal disorders) | 6 | 2
flatulence (Gastrointestinal disorders) | 4 | 2
taste alteration (Gastrointestinal disorders) | 5 | 1
mucositis (functional / symptomatic), oral cavity (Gastrointestinal disorders) | 5 | 0
dry mouth (Gastrointestinal disorders) | 3 | 0
edema: limb (Blood and lymphatic system disorders) | 3 | 0
lipase (Metabolism and nutrition disorders) | 13 | 8
ALT (Metabolism and nutrition disorders) | 6 | 4
amylase (Metabolism and nutrition disorders) | 5 | 4
AST (Metabolism and nutrition disorders) | 4 | 3
hypokalemia (Metabolism and nutrition disorders) | 3 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
metabolic / lab - other (Metabolism and nutrition disorders) | 3 | 1
hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
neuropathy: sensory (Nervous system disorders) | 8 | 7
dizziness (Nervous system disorders) | 6 | 3
pain, head / headache (General disorders) | 10 | 7
pain, joint (General disorders) | 11 | 2
pain, muscle (General disorders) | 6 | 4
pain, extremity - limb (General disorders) | 3 | 1
pain, pain NOS (General disorders) | 3 | 1
pain, other (General disorders) | 3 | 0
voice changes (Respiratory, thoracic and mediastinal disorders) | 3 | 1
rash / desquamation (Skin and subcutaneous tissue disorders) | 19 | 6
pruritus (Skin and subcutaneous tissue disorders) | 12 | 2
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11 | 1
alopecia (Skin and subcutaneous tissue disorders) | 9 | 2
injection site reaction (Skin and subcutaneous tissue disorders) | 6 | 4
dermatology - other (Skin and subcutaneous tissue disorders) | 6 | 4
flushing (Skin and subcutaneous tissue disorders) | 5 | 3
dry skin (Skin and subcutaneous tissue disorders) | 3 | 2
acne (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less